CLINICAL TRIAL: NCT02546193
Title: Outpatient Foley Catheter Compared to Usual Inpatient Care for Cervical Ripening: a Randomized Controlled Trial
Brief Title: Outpatient Foley Catheter Compared to Usual Inpatient Care for Labor Induction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit/accrue adequate numbers of participants within funding period.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vanessa Torbenson, Instructor in Obstetrics-Gynecology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-008988
Record Dates: First submitted 2015-08-14; First posted 2015-09-10 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-05

CONDITIONS: Pregnancy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient Foley catheter (Randomized & Prospective) (Experimental): This arm reflects enrolled women who were (A) randomized to the outpatient Foley catheter group (RCT design) or (B) chose the outpatient Foley catheter group (Modified Prospective study design).
  Participants underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exams the evening before their scheduled induction in the Family Birth Center. A Foley catheter was placed for cervical ripening. After fetal monitoring, they were dismissed to home, to return to the Family Birth Center in the morning for continuation of their labor inductions in the inpatient setting.
  Interventions: Device: Foley catheter
- Inpatient usual care (Randomized & Prospective) (Active Comparator): This arm reflects enrolled women who were (A) randomized to the inpatient usual care group (RCT design) or (B) chose the inpatient usual care group (Modified Prospective study design). No participants in the modified Prospective study design were accrued due to screen failure.
  Participants presented to the Family Birth Center in the evening for their scheduled induction of labor. They underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exam. Cervical ripening commenced with either a Foley catheter or vaginal misoprostol per the discretion of the managing obstetric team. They remained in the inpatient setting throughout their entire labor induction course.
  Interventions: Device: Foley catheter; Drug: Misoprostol

INTERVENTIONS:
Device: Foley catheter — The Foley catheter is a device used to achieve cervical ripening at the start of labor induction. It is a single balloon catheter placed transcervically by a provider, either digitally or using a speculum for visualization. The balloon is placed above the internal os but below the fetal head, amniotic membranes, and placenta and is inflated. In this study, it will be inflated with 60 cc of normal saline and taped to the patient's thigh for traction. Over several hours, the balloon gradually dilates the cervix. The catheter is typically expulsed when the cervix is 3-4 centimeters.
Drug: Misoprostol — Misoprostol is a prostaglandin E1 analogue that is used for cervical ripening during labor induction. A 25 microgram tablet is placed in the vagina by a provider. A new 25 mcg tablet can be used vaginally every 4 hours for up to 6 total doses.
  Arms: Inpatient usual care (Randomized & Prospective)

SUMMARY:
Induction of labor, or causing labor to start before it otherwise starts spontaneously, is sometimes necessary as pregnancy progresses to ensure the safety of both mother and infant. Labor induction often begins with cervical ripening, in which various methods are used to prepare the cervix for contractions and labor. Cervical ripening is beneficial and decreases the need for cesarean section; however, it can be a lengthy process. By tradition, pregnant women are admitted to the hospital at the start of this process and remain inpatient until after the baby is born.

There is increasing interest in allowing the mother to return to her own home during the very first part of this process. She may be more satisfied in a more comfortable environment with her family. Growing scientific evidence supports use of the Foley catheter as an approach to outpatient cervical ripening. The Foley catheter is a safe, effective method that is already used often in the inpatient setting. It does not cause increased health risks for either mother or baby. Previous research studies have shown that it is just as safe and effective when women return to their own homes with a Foley catheter and that women spend less time in the hospital before delivery. More information is needed before this becomes a standard of care. This research study will allow pregnant women to return home for the first night of their labor induction with a Foley catheter in place. In the morning they will return to the hospital and stay until after delivery. They will be compared to a group of women who remain in the hospital for their entire labor induction. The benefits to going home during labor induction may include increasing maternal satisfaction and optimizing the use of resources in the hospital.

DETAILED DESCRIPTION:
This study began as a randomized controlled trial, but due to difficulty enrolling and high screen-failure rates, was modified to a prospective study design allowing participants to choose the arm they wished to participate in at the time of providing informed consent. The intervention group (both designs) was comprised of low risk pregnant women who will have a Foley catheter placed followed by dismissal home with return in the morning for continuation of the labor induction process. The control group consists of women (both designs) who will remain inpatient during the entire cervical ripening phase followed by continuation of the labor induction process in the inpatient setting.

Low risk pregnant women at term will be enrolled in clinic after their providers have recommended induction of labor for a specific indication. They will be educated about induction of labor, the Foley catheter, and the proposed research study. If they would like to participate, they will be consented in the clinic. For the RCT design, a computer-generated randomization would occur on the morning of the planned induction, and the patients will be contacted by phone to inform them of their assigned group. The randomization will be stratified by parity and BMI.

Outpatient Foley catheter group:

If the patient was randomized or chose the intervention group (outpatient Foley), she underwent the following. She will present to the Family Birth Center in the evening at 1900. She will undergo a nonstress test (NST), an ultrasound for fetal presentation and amniotic fluid index, and a cervical exam with calculation of a Bishop score. The patient will be asked if she is having regular, painful contractions, decreased fetal movement, vaginal bleeding, leakage of fluid from the vagina concerning for rupture of membranes, or fevers or chills. A Foley catheter will be placed if the following criteria have been met: the nonstress test is reactive and reassuring (without the presence of ≥ 3 variable decelerations in a 20 minute period, late-appearing decelerations, or any deceleration lasting ≥1 minute), the fetal presentation is cephalic, the amniotic fluid index is 5 centimeters or more, the Bishop score is <6, the cervical dilation is <3 cm, and she has no other clinical characteristics that exclude her from the trial as described in the inclusion/exclusion criteria. A 30 French Foley will be placed either digitally or with speculum assistance. It will be inflated with 60 cc of normal saline and taped to the patient's inner thigh. The fetal heart rate tracing will be monitored for 1 hour after Foley placement. The patient will be sent home if the following criteria are met: the fetal heart rate tracing is reactive and category I; there is no evidence of rupture of membranes, spontaneous labor, or vaginal bleeding more than spotting; and no other exclusion criteria are present. Before discharge, the patient may receive pharmacologic pain relief in the form of one dose of acetaminophen and/or fentanyl.

The patient will be instructed to return to the Family Birth Center at 0700 the following day. She will be given detailed verbal and written instructions of when to contact and return to the Family Birth Center before the morning. She will be provided with the 24 hour direct access line for the Family Birth Center to call with any questions or concerns. If the Foley catheter is expulsed at home, she is to record the time of expulsion. She does not need to return to the Family Birth Center earlier than planned due to expulsion.

When the patient returns in the morning, the induction will be continued at the discretion of the providing obstetric team. The remainder of her care during the first, second, and third stages of labor will be at the discretion of the providing team. The patient will have continuous fetal monitoring. All patients' labor progress will be monitored using a partogram. Cesarean delivery will not be performed for arrest of labor or failed induction unless all criteria have been met as outlined by the Family Birth Center Workgroup protocol made effective 6/2/14.

Inpatient usual care group:

If the patient was randomized or chose the control group (inpatient usual care), she will arrive to the Family Birth Center at 1900 to undergo induction of labor. She will undergo a nonstress test (NST), an ultrasound for fetal presentation and amniotic fluid index, and a cervical exam with calculation of a Bishop score. The patient will be asked if she is having regular, painful contractions, decreased fetal movement, vaginal bleeding, leakage of fluid from the vagina concerning for rupture of membranes, or fevers or chills. She will be included or excluded from the study based on the above information. Induction of labor may proceed at the discretion of the providing obstetric team. Cervical ripening should be performed with either 25 mcg vaginal misoprostol every 4 hours with a maximum of six doses or a 30 Fr Foley catheter filled with 60 cc normal saline. The patient may need both methods during her inpatient stay if her cervix is unfavorable. A Foley catheter will be favored during the cervical ripening phase if there is tachysystole and/or a nonreassuring fetal heart tracing precluding further misoprostol administration, provided the Bishop score is still <6. The remainder of her care during the first, second, and third stages of labor will be at the discretion of the providing team. All patients' labor progress will be monitored using a partogram. Cesarean delivery will not be performed for arrest of labor or failed induction unless all criteria have been met as outlined by the Family Birth Center Workgroup protocol made effective 6/2/14.

Follow up

Each mother was asked to complete a survey before leaving the hospital describing her experience and satisfaction with the cervical ripening process (both study designs. Primary and secondary endpoints will be collected from neonatal and maternal charts through 42 days after the patient's delivery or the date of the patient's final postpartum clinic visit, whichever comes last.

ELIGIBILITY:
Inclusion Criteria

1. Pregnant women at ≥37 weeks gestation by reliable dating criteria as determined by the American College of Obstetricians and Gynecologists (i.e. gestational age supported by one of the following: ultrasound prior to 20 weeks of gestation, fetal heart tones auscultated by Doppler for 30+ weeks, or documented serum or urine pregnancy test 36+ weeks ago)
2. Scheduled induction of labor with indication and timing supported by the Family Birth Center induction of labor guideline entitled "Induction of labor: Indications and Timing"
3. Singleton gestation
4. Cephalic presentation
5. Amniotic fluid index greater than or equal to 5 centimeters
6. Formal prenatal ultrasound documenting the absence of placenta previa
7. Bishop score <6 and cervical dilation <3cm
8. The woman is able to give appropriate consent and has undergone an informed consent process.
9. Maternal age ≥ 18 years old at the time of consent.

Exclusion Criteria

1. New diagnosis requiring immediate hospitalization for monitoring (such as new onset hypertensive disease of pregnancy)
2. Vaginal bleeding
3. Active labor
4. Premature rupture of membranes as determined by positive ferning and as supported by pooling of fluid in the vaginal vault.
5. Uterine tachysystole (>5 contractions in 10 minutes)
6. Nonreassuring fetal heart tracing before or after Foley placement
7. Chorioamnionitis or maternal fever
8. Intrauterine fetal demise
9. Contraindication to vaginal delivery, relative or absolute (i.e. transfundal uterine surgery)
10. Abnormal placentation including a low lying placenta
11. Prior cesarean delivery
12. Intrauterine growth restriction (growth <10th percentile by formal ultrasound)
13. Known fetal anomaly
14. Human immunodeficiency virus, Hepatitis C, or active herpes infection
15. Maternal cardiopulmonary disease requiring cardiac monitoring during labor
16. Pregestational diabetes
17. Rh isoimmunization
18. Non-English speaking
19. Distance from the hospital over 60 minutes by car, unreliable communication via telephone, or unreliable transportation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa E Torbenson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Background] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were enrolled in the outpatient obstetric clinic approximately 2-4 weeks prior to their scheduled induction of labor.
Pre-assignment Details: Women were excluded from the study prior to randomization (the day before their scheduled induction of labor) due to spontaneous onset of labor or other maternal/fetal concern necessitating delivery prior to scheduled induction date.
Groups:
- Outpatient Foley Catheter: Women randomized to the outpatient Foley catheter group underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exams the evening before their scheduled induction in the Family Birth Center. A Foley catheter was placed for cervical ripening. After fetal monitoring, they were dismissed to home, to return to the Family Birth Center in the morning for continuation of their labor inductions in the inpatient setting.
- Inpatient Usual Care: Women randomized to the inpatient usual care group presented to the Family Birth Center in the evening for their scheduled induction of labor. They underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exam. Cervical ripening commenced with either a Foley catheter or vaginal misoprostol per the discretion of the managing obstetric team. They will remained in the inpatient setting throughout their entire labor induction course.
- Prospective Study Outpatient Intervention Group: Women chose the outpatient Foley catheter group underwent basic history review, fetal non-stress testing, ultrasound for presentation and amniotic fluid index, and cervical exams the evening before their scheduled induction in the Family Birth Center. A Foley catheter was placed for cervical ripening. After fetal monitoring, they were dismissed to home, to return to the Family Birth Center in the morning for continuation of their labor inductions in the inpatient setting.
- Prospective Study Inpatient Usual Care Group: Women who chose the inpatient usual care group presented to the Family Birth Center in the evening for their scheduled induction of labor. They underwent basic history review, fetal non-stress testing, ultrasound for presentation and amniotic fluid index, and cervical exam. Cervical ripening commenced with either a Foley catheter or vaginal misoprostol per the discretion of the managing obstetric team. They will remained in the inpatient setting throughout their entire labor induction course.
Period: Overall Study
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care | Prospective Study Outpatient Intervention Group | Prospective Study Inpatient Usual Care Group
Started | 10 | 10 | 2 (Enrolled independently (Prospective study). Not counted in Outpatient Foley Catheter Arm.) | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 6 | 6 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0
Not completed — Not eligible at time of induction | 4 | 6 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Outpatient Foley Catheter (Randomized & Prospective): This arm reflects enrolled women who were (A) randomized to the outpatient Foley catheter group (RCT design) or (B) chose the outpatient Foley catheter group (Modified Prospective study design). NOTE: Baseline data were only collected on women who were accrued, meaning they met eligibility criteria for randomization (RCT design) or met eligibility criteria upon presentation to the Family Birth Center for induction (Modified Prospective study design). No participants in the modified Prospective study design were accrued due to screen failure.
  Participants underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exams the evening before their scheduled induction in the Family Birth Center. A Foley catheter was placed for cervical ripening. After fetal monitoring, they were dismissed to home, to return to the Family Birth Center in the morning for continuation of their labor inductions in the inpatient setting.
- Inpatient Usual Care (Randomized & Prospective): This arm reflects enrolled women who were (A) randomized to the inpatient usual care group (RCT design) or (B) chose the inpatient usual care group (Modified Prospective study design). NOTE: Baseline data were only collected on women who were accrued, meaning they met eligibility criteria for randomization (RCT design) or met eligibility criteria upon presentation to the Family Birth Center for induction (Modified Prospective study design). No participants in the modified Prospective study design were accrued due to screen failure.
  Participants presented to the Family Birth Center in the evening for their scheduled induction of labor. They underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exam. Cervical ripening commenced with either a Foley catheter or vaginal misoprostol per the discretion of the managing obstetric team. They remained in the inpatient setting throughout their entire labor induction course.
- Total: Total of all reporting groups
Arm/Group | Outpatient Foley Catheter (Randomized & Prospective) | Inpatient Usual Care (Randomized & Prospective) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6.3) | 28 (6.0) | 30.5 (0.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pre-delivery Hospitalization Time
Description: The time from when the patient is admitted to the hospital until she delivers her infant and placenta will be recorded. For the outpatient group, this will be measured by adding together the time that the patient spends in the Family Birth Center during Foley placement in the evening with the time she spends inpatient the next day during the rest of her induction until delivery.
Time Frame: Delivery, approximately 16 to 30 hours after admission
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Inpatient Usual Care: Women randomized to the inpatient usual care group presented to the Family Birth Center in the evening for their scheduled induction of labor. They underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exam. Cervical ripening commenced with either a Foley catheter or vaginal misoprostol per the discretion of the managing obstetric team. They remained in the inpatient setting throughout their entire labor induction course.
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
minutes | 1197 (267) | 1398 (264)

2. Secondary Outcome: Mean Score on Maternal Satisfaction Survey
Description: This survey will gauge the mother's experience during her induction with regard to pain, rest, concerns during the induction, satisfaction, and willingness to recommend their particular induction setting (inpatient vs. outpatient). Questions are based on a 1-4 scale, with higher scores indicating greater satisfaction.
Time Frame: Discharge from the hospital, approximately 2-3 days after delivery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
score on a scale | 3.25 (0.5) | 3 (0.8)

3. Secondary Outcome: Number of Participants Per Method of Induction Used
Description: Method of induction: outpatient placement of Foley catheter vs. inpatient usual care induction (medication and/or Foley catheter at time of admission)
Time Frame: End of the third stage of labor, approximately 16 hours after admission
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
Participants | 4 | 4

4. Secondary Outcome: Mean Dose of Medication for Pain Relief
Description: Mean dose of opioid pain medication (Fentanyl) in micrograms
Time Frame: End of the third stage of labor, approximately 16 hours after admission
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
micrograms | 160 (131.9) | 322 (403.9)

5. Secondary Outcome: Mean Time of Delivery
Description: Time from admission to the hospital to delivery of the placenta.
Time Frame: End of the third stage of labor, approximately 16 to 30 hours after admission
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
hours | 19.94 (4.46) | 23.29 (4.39)

6. Secondary Outcome: Number of Participants With Normal Spontaneous Vaginal Delivery
Time Frame: End of the third stage of labor, approximately 16 hours after admission
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
Participants | 3 | 3

7. Secondary Outcome: Mean Estimated Blood Loss at Delivery
Description: Estimated total blood loss at time of delivery in milliliters.
Time Frame: End of the third stage of labor, approximately 16 hours after admission
Measure: Mean (Standard Deviation); unit: milliters
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
milliters | 500 (334.17) | 562.5 (298.26)

8. Secondary Outcome: Number of Participants With Intrapartum Complications
Description: Intrapartum complications defined as intrapartum fever, placental abruption, or chorioamnionitis.
Time Frame: Final postpartum visit, approximately 42 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Postpartum Complications
Description: Postpartum complications defined as postpartum hemorrhage, depression, urinary tract infection, wound infection, endomyometritis, mastitis, pyelonephritis, intra-abdominal infection, deep vein thrombosis, pulmonary thrombosis, cardiac complication, or fever of unknown origin.
Time Frame: Final postpartum visit, approximately 42 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
Participants | 1 | 0

10. Secondary Outcome: Mean Readmission Rate
Description: Defined as readmission to the hospital for any reason within 6 weeks from the date of delivery.
Time Frame: Final postpartum visit, approximately 42 days after delivery
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
readmissions | 0 (0) | 0 (0)

11. Secondary Outcome: Number of Infants Per Gender
Description: Gender defined as male or female.
Time Frame: Neonatal discharge from the hospital, approximately 2-3 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
Participants
  Female | 1 | 2
  Male | 3 | 2

12. Secondary Outcome: Mean Birth Weight
Description: Mean infant birth weight reported in grams.
Time Frame: Neonatal discharge from the hospital, approximately 2-3 days after delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
grams | 3602.5 (184.2) | 3635 (323.2)

13. Secondary Outcome: Mean APGAR Scores
Description: APGAR (Appearance, Pulse, Grimace, Activity, Respiration) Scoring System. 1-10 scale with higher total score indicating better newborn health. Infant mean APGAR score at 5 minutes reported.
Time Frame: Neonatal discharge from the hospital, approximately 2-3 days after delivery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
score on a scale | 9 (0) | 9 (0)

14. Secondary Outcome: Mean Umbilical Cord Blood Gases
Description: Mean infant venous pH reported from complete umbilical cord blood gases.
Time Frame: Neonatal discharge from the hospital, approximately 2-3 days after delivery
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
pH | 7.35 (0.05) | 7.32 (0.04)

15. Secondary Outcome: Number of Infants With Neonatal Morbidity or Mortality, Categorized by Reason.
Description: Any diagnosed neonatal morbid condition or mortality prior to hospital discharge.
Time Frame: Neonatal discharge from the hospital, approximately 2-3 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Foley Catheter | Inpatient Usual Care
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collection period was defined as 42 days following delivery, or the date of the final postpartum visit (typically at 6 weeks), whichever comes last.
Groups:
- Outpatient Foley Catheter (Randomized & Prospective): This arm reflects enrolled women who were (A) randomized to the outpatient Foley catheter group (RCT design) or (B) chose the outpatient Foley catheter group (Modified Prospective study design). NOTE: Adverse events were only collected on women who were accrued, meaning they met eligibility criteria for randomization (RCT design) or met eligibility criteria upon presentation to the Family Birth Center for induction (Modified Prospective study design). No participants in the modified Prospective study design were accrued due to screen failure.
  Participants underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exams the evening before their scheduled induction in the Family Birth Center. A Foley catheter was placed for cervical ripening. After fetal monitoring, they were dismissed to home, to return to the Family Birth Center in the morning for continuation of their labor inductions in the inpatient setting.
- Inpatient Usual Care (Randomized & Prospective): This arm reflects enrolled women who were (A) randomized to the inpatient usual care group (RCT design) or (B) chose the inpatient usual care group (Modified Prospective study design). NOTE: Adverse events were only collected on women who were accrued, meaning they met eligibility criteria for randomization (RCT design) or met eligibility criteria upon presentation to the Family Birth Center for induction (Modified Prospective study design). No participants in the modified Prospective study design were accrued due to screen failure.
  Participants presented to the Family Birth Center in the evening for their scheduled induction of labor. They underwent basic history review, fetal nonstress testing, ultrasound for presentation and amniotic fluid index, and cervical exam. Cervical ripening commenced with either a Foley catheter or vaginal misoprostol per the discretion of the managing obstetric team. They remained in the inpatient setting throughout their entire labor induction course.
Arm/Group | Outpatient Foley Catheter (Randomized & Prospective) | Inpatient Usual Care (Randomized & Prospective)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
No statistical analysis comparing the intervention to usual care was undertaken due to inability to achieve necessary sample size and power required to meaningfully assess the aims and detect statistical effect of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT02546193/Prot_SAP_000.pdf